CLINICAL TRIAL: NCT02195570
Title: Contingency Management for Smoking Cessation in Pregnant Minority Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to identify and recruit eligible participants
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Veronica Accornero, Associate Professor of Clinical Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130654; R34DA031973 (NIH)
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Cigarette Smoking
Keywords: contingency management; smoking cessation; prenatal tobacco exposure; maternal smoking
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QSN with CM (QSN-CM). (Experimental): Women will receive standard of care Quit Smoking Now tobacco education and support plus prize-based contingency management. Their smoking status will be monitored from quit date through 3 months postpartum via carbon monoxide and salivary cotinine levels. Women will earn chances to win prizes each time they test negative for smoking according to biochemical measures.
  Interventions: Other: Quit Smoking Now (QSN); Behavioral: Prize-based Contingency Management (CM)
- QSN Only (Active Comparator): Women receive the standard of care Quit Smoking Now tobacco education and support only. Smoking status will be monitored from quit date through 3 months postpartum via carbon monoxide and salivary cotinine levels. Incentives are given for providing breath and salivary samples but are not contingent on smoking status.
  Interventions: Other: Quit Smoking Now (QSN)

INTERVENTIONS:
Other: Quit Smoking Now (QSN) — The Quit Smoking Now (QSN) program, offered by the Florida Area Health Education Center, was developed based on principles of the Centers for Disease Control and Prevention's "Best Practices for Comprehensive Tobacco Control", and the U.S. Department of Health and Human Services' "Treating Tobacco Use and Dependence Clinical Guidelines" with an emphasis on reaching medically-underserved populations. The QSN curriculum will be delivered in 6 one-hour sessions . Pregnancy-specific session goals and content cover the effects of smoking on the developing fetus, secondhand smoke exposure, the importance of social support, and postpartum relapse.
Behavioral: Prize-based Contingency Management (CM) — Women will earn chances to win prizes for biochemically verified abstinence from tobacco.
  Arms: QSN with CM (QSN-CM).

SUMMARY:
The long-term goal of this research is to reduce tobacco-related disparities in maternal and infant health outcomes by improving smoking cessation and relapse prevention interventions for minority pregnant and postpartum women, who have been significantly underrepresented in smoking cessation research. This study will examine the feasibility and efficacy of a prize-based contingency management approach for increasing smoking cessation and preventing relapse among socioeconomically disadvantaged minority pregnant smokers. First, the intervention will be pretested with 10 pregnant low-income minority smokers and then refined based on acceptability survey and focus group data. Next, a pilot study will be conducted. 60 highly disadvantaged minority women, recruited from the outpatient obstetric clinics at a large teaching hospital, who report daily smoking and who meet other eligibility criteria will be enrolled and randomized to one of two study conditions: 1) Standard Psychoeducational Intervention (6-week, individually-administered, pregnancy-specific Quit Smoking Now curriculum, as currently implemented in the clinic; QSN Only); 2) Standard Psychoeducational Intervention plus Contingency Management (provision of incentives contingent on biochemically-verified abstinence; QSN-CM). Abstinence monitoring via expired carbon monoxide and salivary cotinine levels will occur in both groups beginning on the first quit day and continuing through 3-months postpartum. Only participants in the QSN-CM group will be reinforced for biochemically-verified abstinence with chances to win prizes ranging in value from approximately $1 to $100 ('fishbowl' or 'prize bowl' method). Study outcomes will be assessed through follow-up research exams (delivery and 6-months postpartum) and hospital chart reviews. The primary hypothesis is that that women randomized to the QSN-CM condition will have higher rates of abstinence during pregnancy and postpartum compared to women receiving standard of care alone. Results should advance scientific knowledge regarding effective methods for promoting and maintaining smoking abstinence among pregnant disadvantaged women and provide preliminary feasibility and efficacy data needed to support a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* self-identified daily smoker (at least 1 cigarette/day)
* <28 weeks gestation
* 18 years or older
* resident of Miami-Dade County, Florida
* able to read and speak in English or Spanish
* plans to continue prenatal care with Jackson Health System
* plans to remain in the Miami-Dade County metropolitan area for at least 6 months following delivery.

Exclusion Criteria:

* participation in another smoking cessation intervention within the past year
* use of nicotine replacement therapy (NRT) anytime during pregnancy
* inability to give informed consent
* incarceration
* reported regular use of alcohol (>3 times/week) or marijuana (>weekly); any cocaine or opiates in past year; or a positive toxicology for these drugs.

Study withdrawal will occur in the case of pregnancy termination, fetal demise or by participant request.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Abstinence Duration | (from quit date through 6 months postpartum; assessed up to 52 weeks)
  -duration in days
  --measured by self-report, carbon monoxide, salivary and urine cotinine levels
Abstinence rate (%) | delivery and 6 months postpartum
  * 7-day point prevalence abstinence at delivery and 6 months postpartum defined by no smoking in the 7 days prior to assessment.
  * measured by self-report, carbon monoxide and salivary cotinine levels.
QSN attendance | (6 weeks)
  * cumulative attendance at QSN sessions (1-6 weeks)
  * QSN attendance logs

SECONDARY OUTCOMES:
Smoking reduction | Change (baseline and delivery; baseline and 6 months postpartum)
  -change in the number of cigarettes smoked daily by self-report
Gestational Age | delivery
  * measured in weeks
  * documented through medical chart review
Infant Respiratory Illnesses | 6 months postpartum
  * number of episodes
  * documented through medical chart review
Birth Weight | delivery
  * birth weight measured in grams
  * documented through medical chart review
Neonatal Admissions | delivery
  * duration in days
  * documented through medical chart review

CONTACTS AND LOCATIONS:
Overall Officials: Veronica H Accornero, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States